CLINICAL TRIAL: NCT05899712
Title: Digital Versus Conventional Altered Cast Techniques For Constructing Mandibular Distal Extension Removable Partial Dentures Using Digitally Fabricated Frameworks: A Clinical Comparative Parallel Study of Alveolar Bone Height Changes
Brief Title: Digital Versus Conventional Altered Cast Techniques For Constructing Mandibular Distal Extension Removable Partial Dentures Using Digitally Fabricated Frameworks: Alveolar Bone Height Changes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: A0203023RP
Record Dates: First submitted 2023-06-03; First posted 2023-06-12 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2023-05

CONDITIONS: Denture, Partial, Removable

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Active Comparator): Digitally obtained altered cast for construction of mandibular free end saddle removable partial denture
  Interventions: Other: Removable Partial Denture Construction
- Group B (Active Comparator): Conventionally obtained altered cast for construction of mandibular free end saddle removable partial denture
  Interventions: Other: Removable Partial Denture Construction

INTERVENTIONS:
Other: Removable Partial Denture Construction — Construction of class I Removable partial denture by digital workflow

SUMMARY:
This clinical study compares between digital and conventional altered cast techniques using digitally constructed frameworks in removable partial dentures' construction regarding their effect on bone height changes around abutment teeth and in residual ridge.

ELIGIBILITY:
Inclusion Criteria:

1. All patients having completely edentulous maxilla and class I Kennedy mandible.
2. Sufficient (not less than 15 mm) restorative space must be available (from the mucosa covering the crest of the residual ridge to proposed occlusal plane). This will be detected by a tentative jaw relation.
3. All patients are of angel's class I maxillo-mandibular relationships
4. Abutment teeth must meet certain requirements :

A. Abutment teeth should be healthy with good periodontal and bone support. B. should not show advanced destructions. C. should not show a pronounced degree of mobility or advanced gingival recession.

D. Crown Root Ratio for an abutment is 1:2

Exclusion Criteria:

1. Sever undercuts or concavities on the buccal or lingual sides of the ridge.
2. Systemic diseases that may affect bone changes such as diabetes and osteoporosis.
3. History of radiotherapy in the head and neck region.
4. Crown Root Ratio for an abutment is 1:1.

Ages: 50 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2023-05-15 (Actual); Primary Completion 2025-05-10 (Actual); Study Completion 2025-05-10 (Actual)

PRIMARY OUTCOMES:
Alveolar Bone Height Changes | one year
  Alveolar bone height changes of abutment teeth and residual ridge.

CONTACTS AND LOCATIONS:
Locations (1):
- Mansoura University, Al Mansurah, Dakahlyia, Egypt

IPD SHARING:
Plan to Share IPD: No